CLINICAL TRIAL: NCT02477098
Title: Preoperative Versus Postoperative Ultrasound-guided Rectus Sheath Block for Improving Pain, Sleep Quality and Cytokine Levels of Patients With Open Midline Incisions Undergoing Transabdominal Gynaecological Operation
Brief Title: Preoperative Versus Postoperative Ultrasound-guided Rectus Sheath Block for Sleep Quality and Cytokines of Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Associate professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015110901
Record Dates: First submitted 2015-06-15; First posted 2015-06-22 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Postoperative Pain
Keywords: rectus sheath block; cytokines; sleep
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Postoperative Period

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre RSB (Experimental): patients who receive preoperative rectus sheath block of ropivacaine hydrochloride and receive postoperative rectus sheath block of saline
  Interventions: Drug: preoperative 0.5% ropivacaine hydrochloride preoperative
- Post RSB (Experimental): patients who receive preoperative rectus sheath block of saline and receive postoperative rectus sheath block of Ropivacaine hydrochloride
  Interventions: Drug: postoperative 0.5% Ropivacaine hydrochloride

INTERVENTIONS:
Drug: preoperative 0.5% ropivacaine hydrochloride preoperative — Before surgery (Pre RSB) , a bilateral RSB with ropivacaine hydrochloride will be performed under ultrasound guidance by one anaesthesiologist.At the end of surgery, a bilateral RSB with saline will be performed under ultrasound guidance by one anaesthesiologist.
  Other Names: preoperative rectus sheath block of 0.5% Ropivacaine hydrochloride
  Arms: Pre RSB
Drug: postoperative 0.5% Ropivacaine hydrochloride — Before surgery, a bilateral RSB with saline will be performed under ultrasound guidance by one anaesthesiologist.At the end of surgery, a bilateral RSB with ropivacaine hydrochloride will be performed under ultrasound guidance by one anaesthesiologist.
  Other Names: Rectus sheath block of 0.5% Ropivacaine hydrochloride
  Arms: Post RSB

SUMMARY:
Rectus sheath block (RSB) is used for postoperative pain relief in patients undergoing abdominal surgery with a midline incision. It has proved to be effective in preoperative block, but it has not been previously compared with postoperative block. The aim of the present study is to evaluate postoperative pain, sleep quality and changes in the cytokine levels of patients undergoing gynaecological surgery with RSB performed preoperatively versus postoperatively.

DETAILED DESCRIPTION:
Rectus sheath block (RSB) is used for postoperative pain relief in patients undergoing abdominal surgery with a midline incision. It has proved to be effective in preoperative block, but it has not been previously compared with postoperative block. The aim of the present work is to evaluate the postoperative sleep quality and changes in cytokines of patients undergoing gynaecological operation with RSB preoperatively or postoperatively.

Methods/Design This study is a prospective, randomized, controlled (randomized, parallel group, concealed allocation), double-blinded trial. All patients undergoing transabdominal gynaecological operation will be randomized 1:1 to the treatment intervention with general anaesthesia as an adjunct to RSB preoperatively or postoperatively. The objective of the trial is to evaluate the postoperative sleep quality and changes in cytokines of patients undergoing hysterectomy with RSB preoperatively (n=32) or postoperatively (n=32). All of the patients, irrespective of group allocation, will receive patient-controlled intravenous analgesia with oxycodone.

The primary objective is to compare the interval between leaving the post-anaesthesia care unit and receiving the first PCIA bolus injection on the first postoperative night between patients who receive preoperative versus postoperative RSB. The secondary objectives will be to compare (1) cumulative oxycodone consumption at 24 h after surgery; (2) postoperative sleep quality, as measured using a BIS-Vista monitor during the first night after surgery; and (3) cytokine levels (interleukin-1, interleukin-6, tumour necrosis factor-α and interferon-gamma) during surgery and at 24 and 48 h postoperatively.

ELIGIBILITY:
The inclusion criteria are as follows: (1) an age of 18 to 65 years old; (2) scheduled to undergo elective midline incision transabdominal gynaecological surgery for benign mass; and (3) American Society of Anaesthesiologists (ASA) risk classification I-II.

The exclusion criteria are as follows: (1) patient refusal; (2) known hypersensitivity to the study medication (ropivacaine); (3) long-term use of opioids; (4) liver or renal insufficiency; (5) a history of psychiatric or neurological disease; (6) deafness; (7) previous open surgery; (8) regular use of acetaminophen, nonsteroidal anti-inflammatory drugs, corticosteroids, or antiemetics; and (9) a preoperative Pittsburgh Sleep Quality Index (PSQI) global score of higher than 6

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
the interval between leaving the post-anaesthesia care unit (PACU) and receiving the first PCIA bolus injection | postoperative 24 hours
  The primary objective is to compare the interval between leaving the post-anaesthesia care unit (PACU) and receiving the first PCIA bolus injection on the first postoperative night between patients who receive preoperative RSB and those who receive postoperative RSB.

SECONDARY OUTCOMES:
postoperative pain | postoperative 24 hours
  cumulative oxycodone consumption at 24 h after surgery between patients who receive preoperative versus postoperative RSB
postoperative sleep quality | postoperative 24 hours
  postoperative sleep quality, which will be measured using a BIS-Vista monitor during the first night after surgery
cytokine levels | postoperative 24 and 48 hours
  c)cytokine levels (interleukin-6, tumour necrosis factor-α, interleukin-1 and interferon-gamma ) during the operation and at 24 and 48 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-fei Tan, M.D.,Ph.D, Principal Investigator — First Hospital of China Medical University
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Jin F, Li Z, Tan WF, Ma H, Li XQ, Lu HW. Preoperative versus postoperative ultrasound-guided rectus sheath block for improving pain, sleep quality and cytokine levels in patients with open midline incisions undergoing transabdominal gynecological surgery: a randomized-controlled trial. BMC Anesthesiol. 2018 Feb 9;18(1):19. doi: 10.1186/s12871-018-0485-9. PMID 29426287 (Retraction: PMID 34551704 BMC Anesthesiol. 2021 Sep 23;21(1):230)
- [Derived] Jin F, Li XQ, Tan WF, Ma H, Lu HW. Preoperative versus postoperative ultrasound-guided rectus sheath block for improving pain, sleep quality and cytokine levels of patients with open midline incisions undergoing transabdominal gynaecological operation: study protocol for a randomised controlled trial. Trials. 2015 Dec 10;16:568. doi: 10.1186/s13063-015-1096-0. PMID 26652009